CLINICAL TRIAL: NCT00233155
Title: A Multicenter, Open-Label, Phase 2 Study of NGX-4010 for the Treatment of Neuropathic Pain in Patients With Painful HIV-Associated Neuropathy (HIV-AN) or Postherpetic Neuralgia (PHN)
Brief Title: Study of NGX-4010 for the Treatment of Painful HIV-Associated Neuropathy (HIV-AN) or Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C118
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: Herpes Zoster; Neuralgia; Pain; HIV Infections; Peripheral Nervous System Diseases
Keywords: Analgesics; Capsaicin; Neuropathic pain; Neuropathy; PHN; Shingles
MeSH Terms: conditions — Herpes Zoster; Neuralgia; Pain; HIV Infections; Peripheral Nervous System Diseases

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of NGX-4010 administered at intervals of no less than 12 weeks over 1 year, based on the presence or return of pain, for the treatment of painful HIV-AN and PHN. Participation is limited to former study subjects from previous trials of NGX-4010 at selected sites.

DETAILED DESCRIPTION:
Study C118 is a multicenter, open-label, single-arm study for subjects who successfully completed a previous NGX-4010 study and have not received open-label or blinded NGX-4010 study patches within the 12 weeks prior to study entry. One hundred eligible subjects will receive an initial open-label NGX-4010 study patch application and up to three additional open-label NGX-4010 applications at intervals of no less than 12 weeks, based on the presence or return of pain. Eligible subjects will have moderate to severe neuropathic pain secondary to HIV-AN or PHN, with average pain levels deemed appropriate for further treatment with NGX-4010 as judged by the Investigator.

ELIGIBILITY:
Summary eligibility criteria:

* Subjects must be in good health and have successfully completed a past trial of NGX-4010 with no past occurrence of adverse events that would contraindicate further treatment.
* The time between the last study patch on the previous study and the first study patch on this study must be at least 12 weeks.
* Topical pain medications are exclusionary and require washout prior to study patch application for this study.
* Chronic, nontopical pain medications are allowed but must be stable (not as needed) for a defined period prior to first study patch application.
* Other specific inclusion and exclusion criteria must be met prior to enrollment on the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-08; Study Completion 2006-12

PRIMARY OUTCOMES:
Mean percent change from baseline in "average pain for the past 24 hours" NPRS score (i.e., average of scores during Weeks 12 and 48, compared to baseline).

SECONDARY OUTCOMES:
Proportion of subjects who score 2 or 3 ("Much Improved" or "Very Much Improved") on Patient Impression of Change at Weeks 12, 24, 36 and 48.
Proportion of subjects with significant changes in concomitant pain medication usage during the 2nd through 12th week following study patch application.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Tobias, MD, Study Director — NeurogesX

REFERENCES:
- [Derived] Simpson DM, Gazda S, Brown S, Webster LR, Lu SP, Tobias JK, Vanhove GF; NGX-4010 C118 Study Group. Long-term safety of NGX-4010, a high-concentration capsaicin patch, in patients with peripheral neuropathic pain. J Pain Symptom Manage. 2010 Jun;39(6):1053-64. doi: 10.1016/j.jpainsymman.2009.11.316. PMID 20538187